CLINICAL TRIAL: NCT06536569
Title: A Comparison of the Efficacy of 25g Grieshaber Sharkskin ILM Forceps With Reflex Handle vs Standard 25g Grieshaber ILM Forceps for Internal Limiting Membrane Peeling
Brief Title: Comparison of Efficacy Between ILM Forceps
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Sengi (Industry)
Responsible Party: Principal Investigator, Bryon McKay, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H23-03318
Record Dates: First submitted 2024-07-22; First posted 2024-08-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-07

CONDITIONS: Macular Holes; Epiretinal Membrane
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sharkskin Group (Experimental): 25g Grieshaber Sharkskin ILM Forceps with Reflex Handle
  Interventions: Device: Internal limiting membrane (ILM) Peeling with Sharkskin Forceps
- Standard Group (Active Comparator): 25g Grieshaber standard ILM
  Interventions: Device: Internal limiting membrane (ILM) Peeling with Standard Forceps

INTERVENTIONS:
Device: Internal limiting membrane (ILM) Peeling with Sharkskin Forceps — 25g Grieshaber Sharkskin ILM Forceps with Reflex Handle
  Arms: Sharkskin Group
Device: Internal limiting membrane (ILM) Peeling with Standard Forceps — 25g Grieshaber Standard ILM Forceps
  Arms: Standard Group

SUMMARY:
This study is a Single center, prospective, observational, multi surgeon randomized controlled trial. Subjects will be assessed pre-operatively, operatively and at 1 month postoperatively. Clinical evaluations will include measurement of visual acuity and optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

• 19y and older patients with symptomatic ERM (grade 2-3) or Macular hole (non flap-requiring) for elective ILM peeling surgery.

Exclusion Criteria:

* Co-morbid diabetic retinopathy of any grade.
* Neovascular AMD.
* Previous vitrectomy.
* Previous retinal detachment treated with scleral buckle or pneumatic retinopexy.
* Uncontrolled glaucoma or previous glaucoma surgery.
* Combined phacovitrectomy.
* Macula holes with severity requiring flap.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of attempts to initiate peeling | Surgery (Operative Visit)
  Evaluated by recorded video

SECONDARY OUTCOMES:
Number of handle-ReSite/widefield viewing system lens touches | Surgery (Operative Visit)
  Evaluated by recorded video
Duration of Peel | Surgery (Operative Visit)
  Start to completion of peel
Number of deep retinal grasps | Surgery (Operative Visit)
  Evaluated by recorded video

OTHER OUTCOMES:
Corrected Distance Visual Acuity | 1 Month Postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Bryon McKay, MD, PhD, Principal Investigator — UBC
Locations (1):
- Department of Ophthalmology & Visual Sciences, St Paul's Hospital, Ophthalmology, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No